CLINICAL TRIAL: NCT05017805
Title: Safety and Immunogenicity of COVID-19 Vaccines in Patients With Chronic Liver Disease: A Multi-center Prospective Study
Brief Title: COVID-19 Vaccines in Patients With Chronic Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ky-2021-7-8-1
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-08

CONDITIONS: Liver Disease Chronic
Keywords: Liver Disease Chronic; COVID-19 vaccination
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 doses of vaccine (Experimental): Covid-19 vaccination on day 0, day 25±3, and 6 months after the second dose , respectively，and follow up one and half a year
  Interventions: Biological: COVID-19 Vaccines
- 1 dose of the third vaccination (Experimental): One dose of COVID-19 vaccine and 1 year of follow-up
  Interventions: Biological: COVID-19 Vaccines

INTERVENTIONS:
Biological: COVID-19 Vaccines — One dose (0.5 mL) of coronavirus vaccine was inoculated on day 0 and day 25±3, respectively.

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has caused pandemic since outbreak in 2020.Patients with chronic liver disease (CLD) are at higher risk of mortality and morbidity due to COVID-19. Despite there is a large number of clinical trials of COVID-19 vaccines, only a few participants with chronic liver diseases were included.

DETAILED DESCRIPTION:
This study is a prospective, open-label clinical trial. A total of 300 patients with different cancers including chronic hepatitis, cirrhosis .All of the patients will further accept 18 months follow-up study after vaccination. Safety and immunogenicity will be carefully recorded and detected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Serum ALT and AST are both ≤ 80 U/L.
* HIV and TPHA screening were negative.
* Body temperature ≤37.0℃.

Exclusion Criteria:

* Patients who confirmed the diagnosis of liver cancer by imaging examination (CT/MRI/B scan).
* Patients who are allergic to any component of the vaccine, or have a serious history of vaccine allergy.
* Women who is pregnant, breastfeeding, or planning to be pregnant within 6 months.
* Patients with cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, and severe hypertension can not be well controlled by drugs.
* Patients with severe chronic diseases or diseases can not be controlled well during the progress, such as asthma, diabetes, thyroid disease, etc. Congenital or acquired angioedema / neuroedema.c.
* Patients with urticaria within a year.
* Patients with coagulation disorder.
* Faintng during acupuncture treatment .
* Patients who received other investigational drugs within one month.
* Be receiving anti-TB treatment.
* Other conditions determined by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Safety of coronavirus vaccine | Within 2 months after the first dose of COVID-19 vaccination
  Rate of adverse effects after COVID-19 vaccination
Immunogenicity of coronavirus vaccine | Within 2 months after the first dose of COVID-19 vaccination
  Detected the dynamics and titers of anti-SARS-CoV-2 antibodies

SECONDARY OUTCOMES:
Safety of coronavirus vaccine | Within 18 months after the first dose of COVID-19 vaccination
  Rate of adverse effects after COVID-19 vaccination
Immunogenicity of coronavirus vaccine | Within 18 months after the first dose of COVID-19 vaccination
  Detected the dynamics and titers of anti-SARS-CoV-2 antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Cornberg M, Buti M, Eberhardt CS, Grossi PA, Shouval D. EASL position paper on the use of COVID-19 vaccines in patients with chronic liver diseases, hepatobiliary cancer and liver transplant recipients. J Hepatol. 2021 Apr;74(4):944-951. doi: 10.1016/j.jhep.2021.01.032. Epub 2021 Feb 6. PMID 33563499
- [Result] Fix OK, Blumberg EA, Chang KM, Chu J, Chung RT, Goacher EK, Hameed B, Kaul DR, Kulik LM, Kwok RM, McGuire BM, Mulligan DC, Price JC, Reau NS, Reddy KR, Reynolds A, Rosen HR, Russo MW, Schilsky ML, Verna EC, Ward JW, Fontana RJ; AASLD COVID-19 Vaccine Working Group. American Association for the Study of Liver Diseases Expert Panel Consensus Statement: Vaccines to Prevent Coronavirus Disease 2019 Infection in Patients With Liver Disease. Hepatology. 2021 Aug;74(2):1049-1064. doi: 10.1002/hep.31751. PMID 33577086